CLINICAL TRIAL: NCT02274532
Title: Myoelectric SoftHand Pro to Improve Prosthetic Function for People With Below-elbow Amputations: A Feasibility Study
Acronym: SoftHand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen L. Andrews, M.D. (Other)
Collaborators: Arizona State University (Other); University of Pisa (Other)
Responsible Party: Sponsor-Investigator, Karen L. Andrews, M.D., Associate Professor of Physical Medicine & Rehab, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 13-008649
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Upper Limb Amputation Below Elbow (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Experimental): Testing will include self-report questionnaires, assessments of activities of daily living (ADL) by an occupational therapist, and biomechanical measures of forces applied to objects and motion of the upper limb collected during commonly-performed tasks. Motion will be recorded using sensors that are attached to the arm and SoftHand. During each session, videos will be obtained of the subjects performing tasks. The experimental data collections are organized into 5 Sessions, which will take place over the course of 1 week, scheduled by the subject's availability, with the option with patients for a 1-week period of take-home testing and associated pre- and post-assessments.
  Interventions: Device: SoftHand
- Control (Other): Testing will include self-report questionnaires, assessments of activities of daily living (ADL) by an occupational therapist, and biomechanical measures of forces applied to objects and motion of the upper limb collected during commonly-performed tasks. Motion will be recorded using sensors that are attached to the arm and SoftHand. During each session, videos will be obtained of the subjects performing tasks. The experimental data collections are organized into 4 Sessions, which will take place over the course of 1 week, scheduled by the subject's availability. Control subjects will participate in two sessions, including a pre- and post-training assessments.
  Interventions: Device: SoftHand

INTERVENTIONS:
Device: SoftHand — Biomechanical, ADL, and functional testing.
  Other Names: SH; SHpro

SUMMARY:
A study to investigate the hypothesis that a Pisa/IIT Robotic SoftHand Pro converted to a prosthetic terminal device will enhance the performance of people with limb loss in a wider range of daily living tasks than allowed by today's commercially available prosthetic hands, and will exceed established benchmarks for activities of daily living (ADL).

DETAILED DESCRIPTION:
Preliminary data suggest that the SoftHand Pro (SHpro) is extremely versatile and can be used to grasp and manipulate common objects. We will perform extensive testing of the myoelectric SHpro by asking subjects to perform a wide variety of ADL tasks in a structured environment onsite at Mayo Clinic Rochester. These data will be used by the Mayo Clinic, ASU, and the IIT research teams to modify the SHpro design to adapt it for use by people with amputations while focusing on the SHpro socket design, surface electromyography (EMG)-based control (typically used in commercially available prostheses today).

We will quantify the ability of patients with below-elbow amputation to perform the above tasks using the prosthetic terminal device version of the SHpro. We hypothesize that people with amputations will learn to use the SHpro and perform grasp and manipulation tasks to a greater level than that allowed by their current terminal devices.

The long-term objectives of this exploratory study are to design and build a low-cost, high-performance prosthetic hand terminal device that will be accepted by patients with below-elbow amputation and allow them to perform a wider range of ADL tasks than allowed by today's commercially available prostheses. The data collected through the proposed studies will provide an important foundation for optimizing the design of the SHpro for future testing on a large number of people with limb loss. Future studies will also assess the extent to which the SHpro's functionality and acceptance might benefit from embedding additional synergistic hand motion patterns in the SHpro.

ELIGIBILITY:
Inclusion Criteria:

1) Subjects > 18 years of age.

Exclusion Criteria:

1. Patients with an amputation for less than 6 months.
2. Patients who have been fit and trained to use a prothesis but chose not to do so.
3. Clinical history of brachial plexopathy, cervical radiculopathy or polyneuropathy and persistent weakness.

5) Visual problems that would interfere with our grasp task.

6) Co-existing central nervous system disease (e.g., multiple sclerosis, motor neuron disease, myasthenia gravis, Parkinson's disease, dystonia) that would interfere with our grasp task

7) Significant spasticity/rigidity as assessed through range of motion testing that would interfere with our grasp task.

8) Active psychiatric illness.

9) Cognitive impairments which would interfere with following study instructions and filling out surveys (at the investigator's discretion).

10) Use of medications that might affect sensory and/or motor functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
Functional assessments | 1 week
  DASH score, the Jebsen Taylor Test of Hand Function, and biomechanical measures (including total grip force, load force sharing between the thumb and finger(s), time to peak grip force, and net torque exerted by the subject at object lift onset).

SECONDARY OUTCOMES:
ADL tests | 1 week
  The AM-ULA ADL assessment will be used as secondary outcome measures to identify specific grasping tasks or task component(s) that a control or people with amputations subject might have difficulty performing.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Andrews, M.D., Principal Investigator — Mayo Clinic